CLINICAL TRIAL: NCT01176747
Title: In-vivo Deposition Measurement of Beclometasone and Formoterol After Inhalation of a Single Dose of the Combination BDP Plus Formoterol NEXT DPI in Healthy Volunteers, Asthmatic and COPD Patients.
Brief Title: Lung Deposition of the BDP/Formoterol Combination Administered Via the NEXT DPI in Healthy, Asthmatic and COPD Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Marisa Minetti, website administrator, Chiesi Farmaceutici S.p.A.
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCD-0815-PR-0011; 2009-010267-17 (EudraCT Number)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BDP/formoterol NEXT DPI (Experimental): Radiolabelled BDP/formoterol 100/6 µg dry powder administered via the NEXT inhaler
  Interventions: Drug: BDP/formoterol NEXT DPI

INTERVENTIONS:
Drug: BDP/formoterol NEXT DPI — Single inhalation of radiolabelled BDP/formoterol 100/6 µg NEXT DPI (4 puffs giving a total dose of 400 µg BDP + 24 µg formoterol)
  Other Names: CHF 1535 NEXT DPI

SUMMARY:
The purpose of this study is to investigate the lung deposition and distribution pattern of Beclometasone and Formoterol using a gamma-scintigraphic technique after inhalation of a single dose of 99mTc-radiolabelled BDP/formoterol fixed combination administered Via the NEXT DPI in healthy volunteers, asthmatic and COPD patients. Additionally, the systemic exposures to formoterol, BDP and its monopropionate metabolite (B17MP) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Males and females aged 18-65 years;
* Body Mass Index (BMI) between 18.0 and 28.0 kg/m2;
* Non- or ex-smokers who smoked < 5 pack years and stopped smoking > 1 year;
* Normal blood pressure and heart rate;
* Normal electrocardiogram (ECG,12 lead);
* Normal laboratory tests;

Patients with Asthma:

* Males and females aged 21-65 years;
* BMI between 18.0 and 28.0 kg/m2;
* Non- or ex-smokers who smoked < 5 pack years and stopped smoking > 1 year;
* Normal blood pressure and heart rate;
* Normal ECG (12 lead);
* FEV1 ≥ 30% and < 80% of predicted according to European Coal and Steel Community values (ECSC)
* Reversibility of FEV1 ≥ 12% and at least 200 ml of the initial value 15 minutes after inhalation of 200 µg Salbutamol;

Patients with COPD:

* Males and females aged 40 - 70 years
* BMI between 18.0 and 30.0 kg/m2;
* Normal blood pressure and heart rate;
* Normal ECG (12 lead);
* Stable COPD within the past 4 weeks;
* Post bronchodilator FEV1 between 30% and 50% predicted values (ECSC);
* Post bronchodilator FEV1/FVC < 0.70 (absolute value);
* Minimum smoking history of 10 pack-years;

Exclusion Criteria:

All subjects:

* Blood donation or blood loss in the previous 8 weeks;
* Positive HIV1 or HIV2 serology;
* Positive acute or chronic Hepatitis B or Hepatitis C;
* Unsuitable veins for repeated venipuncture;
* Female patients: pregnant, positive pregnancy test, lactating mother or lack of efficient contraception.
* History of substance abuse or positive urine drug screen;
* Abnormal laboratory values suggesting an unknown disease and requiring further clinical investigation;
* Uncontrolled cardiac, hepatic, renal, gastrointestinal, endocrine, metabolic, neurologic, or psychiatric clinically significant disorder;
* Participation in another clinical trial in the previous 8 weeks; participation in study using radioactive material within 1 calendar year;
* Known sensitivity to Formoterol or Beclometasone or any of the excipients;
* Concomitant severe diseases or diseases which are contra indications for the use of inhaled Beta-2-agonist or steroids;
* Use of any prescription drug for which concomitant beta-agonist or steroid administration are contraindicated;
* Recent relevant infectious disease (less than two months);
* Flu vaccination or other vaccination within 4 weeks prior to the screening visit;

Additional exclusion criteria for healthy volunteers:

* Lung function measurements outside normal limits (normal values: FEV1/FVC > 0.70 and FEV1 and FVC > 80% for the ECSC predicted values);

Additional exclusion criteria for patients with Asthma:

* Use of systemic steroids 4 weeks prior to inclusion (injectable depot steroids 6 weeks) or more than 3 periods during the last 6 months;
* Life-threatening/unstable respiratory status within the previous 30 days;
* Requirement of supplemental oxygen therapy;
* Change in dose or type of any medications for asthma within 4 weeks prior to the screening visit;
* Asthma exacerbation within the 4 weeks prior to inclusion.

Additional exclusion criteria for patients with COPD:

* Use of systemic steroids 4 weeks prior to inclusion (injectable depot steroids 6 weeks) or more than 3 periods during the last 6 months;
* Life-threatening/unstable respiratory status within the previous 30 days;
* Requirement of supplemental oxygen therapy;
* Change in dose or type of any medications for COPD within 4 weeks prior to the screening visit;
* COPD exacerbation within the 4 weeks prior to inclusion;
* History of asthma or any chronic respiratory diseases other than COPD.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Lung deposition of BDP and Formoterol (expressed as % of emitted dose) when inhaled using the NEXT dry powder inhaler | Immediately after dosing
  Calculated using the individual Gamma camera images and the regions of interest defined from the 81mKrypton-ventilation scan.

SECONDARY OUTCOMES:
Distribution of lung deposition | Immediately after dosing
Extrathoracic deposition | Immediately after dosing
Exhaled activity | Immediately after dosing
Plasma pharmacokinetics of formoterol, BDP and its monopropionate metabolite (B17MP) | over 24 h post dose
Lung function parameters | over 24 h post dose

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Meyer, MD, Principal Investigator — Inamed Research GmbH & Co. KG
Locations (1):
- Inamed Research GmbH & Co. KG, Gauting, Germany

REFERENCES:
- [Result] Virchow JC, Poli G, Herpich C, Kietzig C, Ehlich H, Braeutigam D, Sommerer K, Haussermann S, Mariotti F. Lung Deposition of the Dry Powder Fixed Combination Beclometasone Dipropionate Plus Formoterol Fumarate Using NEXThaler(R) Device in Healthy Subjects, Asthmatic Patients, and COPD Patients. J Aerosol Med Pulm Drug Deliv. 2018 Oct;31(5):269-280. doi: 10.1089/jamp.2016.1359. Epub 2018 Jul 10. PMID 29989511
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2009-010267-17
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-0815-PR-0011.pdf